CLINICAL TRIAL: NCT02376192
Title: Maternal Microcirculation & SDF Imaging: A Novel Assessment of the Microcirculation During Cesarean Delivery With Spinal Anesthesia and the Impact of Phenylephrine Prophylaxis to Prevent Spinal Anesthesia-induced Hypotension.
Brief Title: Maternal Microcirculation & SDF Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Director of Medical Research, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IWK1010276
Record Dates: First submitted 2014-09-03; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Pregnancy
Keywords: Microcirculation; Sidestream Dark Field (SDF) Imaging; Spinal Anesthesia; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bolus Phenylephrine/Ephedrine Treatment' (Experimental): Initial MicroScan® (Microvision Medical) SDF measurement are recorded in the obstetric preoperative area within two hours prior to administration of spinal anesthesia. In the operating room participants will receive a standard spinal anesthetic (hyperbaric bupivacaine, fentanyl and preservative free morphine) followed by a second comparative MicroScan® (Microvision Medical) SDF measurement within 10 minutes of initiation of spinal anesthetic. Participants who experience hypotension will receive bolus phenylephrine and/or ephedrine treatment as needed.
  Interventions: Device: Initial MicroScan® (Microvision Medical) SDF Measurement; Drug: Spinal Anesthesia- Bupivacaine; Device: Comparative MicroScan® (Microvision Medical) SDF Measurement; Drug: Bolus Phenylephrine/Ephedrine Treatment
- Phenylephrine Infusion Group (Experimental): Initial MicroScan® (Microvision Medical) SDF measurement are recorded in the obstetric preoperative area within two hours prior to administration of spinal anesthesia. In the operating room participants will receive a standard spinal anesthetic (hyperbaric bupivacaine, fentanyl and preservative free morphine) followed by a second comparative MicroScan® (Microvision Medical) SDF measurement within 10 minutes of initiation of spinal anesthetic. Participants will have an infusion of phenylephrine started immediately following the induction of spinal anesthesia for prevention of hypotension.
  Interventions: Device: Initial MicroScan® (Microvision Medical) SDF Measurement; Drug: Spinal Anesthesia- Bupivacaine; Device: Comparative MicroScan® (Microvision Medical) SDF Measurement; Drug: Phenylephrine Infusion

INTERVENTIONS:
Device: Initial MicroScan® (Microvision Medical) SDF Measurement — Initial SDF measurements are recorded in the obstetric preoperative area within two hours prior to administration of spinal anesthesia.
Drug: Spinal Anesthesia- Bupivacaine — The spinal anesthetic technique is standardized. In the operating room spinal anesthesia will be administered with the L2-L5 interspaces in the sitting position using 12 mg of hyperbaric bupivacaine with 15 mcg of fentanyl and 150 mcg of preservative free morphine.
Device: Comparative MicroScan® (Microvision Medical) SDF Measurement — A second comparative SDF measurement be recorded within 10 minutes after induction of spinal anesthesia.
Drug: Bolus Phenylephrine/Ephedrine Treatment — Participants who experience hypotension following induction of spinal anesthesia will be treated with a bolus of phenylephrine and/or ephedrine as needed.
  Arms: Bolus Phenylephrine/Ephedrine Treatment'
Drug: Phenylephrine Infusion — Participants will have an infusion of phenylephrine started immediately following the induction of spinal anesthesia for prevention of hypotension.
  Arms: Phenylephrine Infusion Group

SUMMARY:
This is a study of pregnant women undergoing a cesarean delivery. It will compare their microcirculation before and after the anesthetic. Microcirculation means blood flow to the extremely small blood vessels in the body. It will also look at the differences in microcirculation of participants who receive an infusion of phenylephrine compared to participants who don't. The investigators hypothesize that spinal anesthesia will reduce the vascular density and proportion of perfused vessels.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status I-II (ASA I - Healthy, ASA II - mild and controlled systemic disease)
* Singleton pregnancies
* 36-42 weeks gestation
* Non-labouring
* Scheduled cesarean delivery
* English speaking
* Age 18-45 years

Exclusion Criteria:

* Cardiovascular disease
* Hypertensive disease of pregnancy (i.e. mild & severe preeclampsia)
* Allergy to phenylephrine, or any other standardized medication
* Obesity (BMI > 35 kg/m2)
* Diabetes Mellitus type 1
* Smoker
* Coffee/Caffeine intake within 6 hours of SDF measurement

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Microvascular Flow Index (MFI) | Immediately prior to, and within 10 minutes of induction of spinal anesthesia
  The change in MFI of participants; measured immediately prior to, and within 10 minutes following the induction of spinal anesthesia

SECONDARY OUTCOMES:
Microvascular Flow Index (MFI) | Immediately prior to, and within 10 minutes of induction of spinal anesthesia
  The difference between the MFI measured within 10 minutes following the induction of spinal anesthesia in participants who receive phenylephrine via a continuous infusion for the prevention of spinal anesthesia-induced hypotension compared to those who may receive phenylephrine boluses for treatment of spinal anesthesia-induced hypotension.

OTHER OUTCOMES:
Total Vessel Density (TVD) | Immediately prior to, and within 10 minutes of induction of spinal anesthesia
Perfused Vessel Density (PVD) | Immediately prior to, and within 10 minutes of induction of spinal anesthesia
Proportion of perfused vessels (PPV) | Immediately prior to, and within 10 minutes of induction of spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD FRCPC, Principal Investigator — IWK Health Centre, Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] George RB, DesRoches J, Abdo I, Lehmann C. Maternal microcirculation and sidestream dark field imaging: a prospective assessment of the association between labour pain and analgesia on the microcirculation of pregnant women. Clin Hemorheol Microcirc. 2015;60(4):389-95. doi: 10.3233/CH-141851. PMID 24934438
- [Background] Abdo I, George RB, Farrag M, Cerny V, Lehmann C. Microcirculation in pregnancy. Physiol Res. 2014;63(4):395-408. doi: 10.33549/physiolres.932511. Epub 2014 Apr 3. PMID 24702490
- [Background] George RB, Munro A, Abdo I, McKeen DM, Lehmann C. An observational assessment of the sublingual microcirculation of pregnant and non-pregnant women. Int J Obstet Anesth. 2014 Feb;23(1):23-8. doi: 10.1016/j.ijoa.2013.08.013. Epub 2013 Sep 8. PMID 24342223
- [Background] Lehmann Ch, Abdo I, Kern H, Maddison L, Pavlovic D, Sharawi N, Starkopf J, Hall R, Johnson P, Williams L, Cerny V; MiDAS (Microcirculation Diagnostics and Applied Studies) group. Clinical evaluation of the intestinal microcirculation using sidestream dark field imaging--recommendations of a round table meeting. Clin Hemorheol Microcirc. 2014;57(2):137-46. doi: 10.3233/CH-141810. PMID 24448730